CLINICAL TRIAL: NCT03702608
Title: Prospective, Multi-center, Single-arm, Open-label Clinical Trial, to Further Assess the Safety and Efficacy of Long (38 mm) Ridaforolimus Eluting Stent - EluNIR
Brief Title: BIONICS 38 mm Trial EluNIR Ridaforolimus Eluting Coronary Stent System (EluNIR) In Coronary Stenosis Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EluNIR-004
Record Dates: First submitted 2018-09-02; First posted 2018-10-11 (Actual); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-05

CONDITIONS: Coronary Stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- EluNIR 38mm (Other)
  Interventions: Combination Product: EluNIR Ridaforolimus Eluting Coronary Stent System

INTERVENTIONS:
Combination Product: EluNIR Ridaforolimus Eluting Coronary Stent System — The EluNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising of:
  * Stent - a mounted Cobalt Chromium (CoCr) alloy based stent - 38 mm length and 2.75mm, 3.0 mm, 3.5mm, 4.0mm diameter
  * Delivery System - Rapid Exchange (RX) Coronary System
  * Polymer matrix coating - (PBMA) and CarboSil®
  * Ridaforolimus drug

SUMMARY:
This is a prospective, multi-center, single-arm, open-label clinical trial. Clinical follow-up will be performed at 30 days. Follow-up by phone will be performed at 6 months, and 1 year after the procedure. Study Objective is to further assess the safety and efficacy of long (38 mm) Ridaforolimus Eluting Stent - EluNIR.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria:

  1. Age ≥ 18 years.
  2. Patient with an indication for PCI including angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present), NSTEMI, or recent STEMI. For STEMI the time of presentation to the first treating hospital, whether a transfer facility or the study hospital, must be >24 hours prior to enrollment and enzyme levels (CK-MB or Troponin) demonstrating that either or both enzyme levels have peaked.
  3. An attempt (whether successful or not) was made to implant a 38 mm EluNIR stent (Stent was advanced beyond the guiding catheter).
  4. Non-target vessel PCI are allowed prior to the screening for eligibility depending on the time interval and conditions as follows:

     1. During Baseline Procedure:

        PCI of non-target vessels performed during the baseline procedure itself immediately prior to screening for eligibility, if successful and uncomplicated defined as: <50% visually estimated residual diameter stenosis, TIMI Grade 3 flow, no dissection ≥ NHLBI type C, no perforation, no persistent ST segment changes, no prolonged chest pain, no TIMI major or BARC type 3 bleeding.
     2. Less than 24 hours prior to Baseline Procedure:

     Not allowed (see exclusion criteria #2). c. 24 hours-30 days prior to Baseline Procedure: i. PCI of non-target vessels 24 hours to 30 days prior to the baseline procedure if successful and uncomplicated as defined above.

     ii. In addition, in cases where non-target lesion PCI has occurred 24-72 hours prior to the baseline procedure, at least 2 sets of cardiac biomarkers must have been drawn at least 6 and 12 hours after the non-target vessel PCI.

     iii. If cardiac biomarkers are initially elevated above the local laboratory upper limit of normal, serial measurements must demonstrate that the biomarkers are falling.

     d. Over 30 days prior to Baseline Procedure: PCI of non-target vessels performed greater than 30 days prior to baseline procedure whether or not successful and uncomplicated.
  5. Patient or legal guardian is willing and able to provide informed written consent and comply with follow-up visits and testing schedule.

     Angiographic inclusion criteria (visual estimate):
  6. Target lesion(s) must be located in a native coronary artery or bypass graft conduit with visually estimated diameter of ≥2.75 mm to ≤4.25 mm.
  7. Complex lesions are allowed including calcified lesions (lesion preparation with scoring/cutting and rotational atherectomy are allowed), presence of thrombus, CTO, bifurcation lesions, ostial RCA lesions, tortuous lesions, bare metal stent restenotic lesions, protected left main lesions, and saphenous vein graft lesions.
  8. Overlapping stents are allowed as long as the first stent implanted is the EluNIR 38 mm long stent

Exclusion Criteria:

* General Exclusion Criteria:

  1. STEMI within 24 hours of initial time of presentation to the first treating hospital, whether at a transfer facility or the study hospital or in whom enzyme levels (either CK-MB or Troponin) have not peaked.
  2. PCI within the 24 hours preceding the baseline procedure.
  3. Non-target lesion PCI in the target vessel within 12 months of the baseline procedure.
  4. History of stent thrombosis.
  5. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including IABP.
  6. Subject is intubated.
  7. Known LVEF <30%.
  8. Relative or absolute contraindication to DAPT for 6 months in non-ACS patients and 12 months in ACS patients (including planned surgeries that cannot be delayed, or subject is indicated for chronic oral anticoagulant treatment).
  9. eGFR <30 mL/min
  10. Hemoglobin <10 g/dL.
  11. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
  12. White blood cell (WBC) count <3,000 cells/mm3.
  13. Clinically significant liver disease.
  14. Active peptic ulcer or active bleeding from any site.
  15. Bleeding from any site within the prior 8 weeks requiring active medical or surgical attention.
  16. If femoral access is planned, significant peripheral arterial disease which precludes safe insertion of a 6F sheath.
  17. History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
  18. Cerebrovascular accident or transient ischemic attack within the past 6 months, or any permanent neurologic defect attributed to CVA.
  19. Known allergy to the study stent components cobalt, nickel, chromium, molybdenum, Carbosil®, PBMA, or limus drugs (ridaforolimus, zotarolimus, tacrolimus, sirolimus, everolimus, or similar drugs or any other analogue or derivative or similar compounds).
  20. Known allergy to protocol-required concomitant medications such as aspirin, or DAPT (clopidogrel, prasugrel, ticagrelor), or heparin and bivalirudin, or iodinated contrast that cannot be adequately pre-medicated.
  21. Any co-morbid condition that may cause non-compliance with the protocol (e.g. dementia, substance abuse, etc.) or reduced life expectancy to <24 months (e.g. cancer, severe heart failure, severe lung disease).
  22. Patient is participating in or plans to participate in any other investigational drug or device clinical trial that has not reached its primary endpoint.
  23. Women who are pregnant or breastfeeding.
  24. Women who intend to become pregnant within 12 months after the baseline procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the baseline procedure).
  25. Patient has received an organ transplant or is on a waiting list for an organ transplant.
  26. Patient is receiving or scheduled to receive chemotherapy within 30 days before or any time after the baseline procedure.
  27. Patient is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease (e.g., HIV). Corticosteroids are allowed.

      Angiographic Exclusion Criteria (visual estimate):
  28. Unprotected left main lesions ≥30%, or planned left main intervention.
  29. Bifurcation lesions with planned dual stent implantation.
  30. Stenting of lesions due to DES restenosis.
  31. Occlusive thrombus and/or a thrombus requiring thrombectomy in a target vessel
  32. Another lesion in a target or non-target vessel (including all side branches) is present that requires or has a high probability of requiring PCI within 12 months after the baseline procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medinol LTD, Tel Aviv, Israel

REFERENCES:
- [Derived] Jonas M, Ben-Yehuda O, Banai S, Segev A, Danenberg H, Assali A, Tuvali O, Haberman D, Chernin G. Percutaneous coronary intervention with ridaforolimus-eluting stents in long lesions: the BIONICS 38 mm prospective trial. Coron Artery Dis. 2023 Sep 1;34(6):410-414. doi: 10.1097/MCA.0000000000001264. Epub 2023 Jul 4. PMID 37471280

RESULTS

PARTICIPANT FLOW:
Groups:
- EluNIR 38mm: Patients received the EluNIR Ridaforolimus Eluting Coronary Stent System: The EluNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising of:
  * Stent - a mounted Cobalt Chromium (CoCr) alloy based stent - 38 mm length and 2.75mm, 3.0 mm, 3.5mm, 4.0mm diameter
  * Delivery System - Rapid Exchange (RX) Coronary System
  * Polymer matrix coating - (PBMA) and CarboSil®
  * Ridaforolimus drug
Period: Overall Study
Arm/Group | EluNIR 38mm
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with an indication for PCI including angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present), NSTEMI, or recent STEMI.
Arm/Group | EluNIR 38mm
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Israel | 50

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint: Device Success
Description: Device success is defined as achievement of a final in-stent residual diameter stenosis of <50% (by QCA), using the assigned device only and without a device malfunction.
Time Frame: 30 day
Measure: Count of Participants; unit: Participants
Arm/Group | EluNIR 38mm
Number analyzed (Participants) | 50
Participants | 44

2. Primary Outcome: Primary Endpoint: No 30 Day MACE (Major Adverse Cardiac Events)
Description: No 30 day MACE: MACE (Major Adverse Cardiac Events) is defined as the composite of cardiac death, any MI, or ischemia-driven TLR.
Time Frame: 30 Day
Measure: Count of Participants; unit: Participants
Arm/Group | EluNIR 38mm
Number analyzed (Participants) | 50
Participants | 44

ADVERSE EVENTS:
Time Frame: The Investigator monitored the occurrence of adverse events or device deficiencies for each subject during the whole course of the trial- baseline and post procedure, 30 days, 6 months and 1 year visits.
Arm/Group | EluNIR 38mm
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 5/49
Other Adverse Events (participants affected / at risk) | 15/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EluNIR 38mm (N=49)
General disorders and administration site conditions (General disorders) | 2
Infections and infestations (Infections and infestations) | 2
Cardiac disorders (Cardiac disorders) | 4
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1
Vascular disorders (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EluNIR 38mm (N=49)
Cardiac disorders (Cardiac disorders) | 7
General disorders and administration site conditions (General disorders) | 4
Infections and infestations (Infections and infestations) | 3
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1
Investigations (Investigations) | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1
Psychiatric disorders (Psychiatric disorders) | 1
Renal and urinary disorders (Renal and urinary disorders) | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1
Vascular disorders (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT03702608/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT03702608/SAP_002.pdf